CLINICAL TRIAL: NCT00378313
Title: A Phase 2 Study of Neoadjuvant Chemotherapy With Gemcitabine, Epirubicin and Paclitaxel (Taxol)[GET] in Locally Advanced Breast Cancer
Brief Title: A Study of Gemcitabine, Epirubicin, and Paclitaxel Combination Chemotherapy Given Before Surgery to Patients With Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP-FB-GE-001
Record Dates: First submitted 2006-09-07; First posted 2006-09-19 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IV Breast Cancer; Breast Cancer; Locally Advanced
Keywords: NSABP; gemcitabine; epirubicin; paclitaxel; Taxol; breast cancer; neoadjuvant chemotherapy; primary chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Epirubicin; Paclitaxel

INTERVENTIONS:
Drug: gemcitabine, epirubicin, paclitaxel

SUMMARY:
The primary purpose of this study is to determine whether locally advanced breast cancer responds (by shrinking, by not progressing or by being destroyed) to combined chemotherapy (gemcitabine, epirubicin and paclitaxel) given before surgery to patients with locally advanced breast cancer. This study will also evaluate the toxicity of the chemotherapy combination to patients and will determine survival and progression-free survival 2 years after treatment. Also, the study will look at whether there are molecular and genetic changes in the tumor tissue that match the tumor's response to the chemotherapy.

DETAILED DESCRIPTION:
Primary chemotherapy has had an established role in locally advanced breast cancer. Studies have shown that the combination of chemotherapeutic agents is superior to single therapeutic agent in overall response rate and progression free survival. The inclusion of the most active drugs in combination regimens can improve the percentage of patients achieving a pathological complete response (pCR). The chemotherapy agents gemcitabine, epirubicin, and paclitaxel have been used individually to treat breast cancer. While use of the combination of these three drugs has been studied in the metastatic setting, the combination has not been evaluated in locally advanced disease. In this study the combination of the three agents gemcitabine, epirubicin, and paclitaxel [Taxol] will be administered to patients with locally advanced breast cancer prior to surgery; pathologic response will be determined at the time of surgery. The main objective of this study is to determine the pathological response rate for these patients. Also because prior studies have suggested that only a specific subset of tumors responds to a specific chemotherapeutic agent and that this subset is determined by the gene expression profile of each tumor, preoperative therapy protocols such as this provide an ideal setting to identify gene expression pattern and gene copy number changes that may predict response to a specific therapy using high-throughput assay methods and RNAlater. Therefore, this study will also look at the feasibility of tissue collection and analysis in identifying predictive markers of complete pathological response.

ELIGIBILITY:
Inclusion criteria:

* Females only
* Consent for the collection of biopsy tissue in RNAlater solution
* Biopsy specimens that were obtained by core biopsy or incisional biopsy and placed in RNAlater solution
* Breast cancer that is:

  * unilateral
  * diagnosed histologically as invasive breast cancer without evidence of metastatic disease (except for stage IV with positive supraclavicular nodes only)
  * stage IIB, IIIA (T0-3N2), IIIB (T4N0-3 or T0-3N3), or IV (by involvement of positive supraclavicular nodes only). (Patients with clinical evidence of inflammatory breast cancer or superficial lesions must have a measurable mass in the breast or lymph nodes.)
  * measurable by physical exam, mammography, sonogram, CT scan, MRI, or x-ray
* Evidence of adequate organ function (liver, bone marrow, kidney)
* Ability to perform an adequate level of physical activity (Zubrod scale 0, 1, or 2)
* Life expectancy of at least 10 years
* Childbearing potential terminated by surgery, radiation, or menopause, or attenuated by use of an effective non-hormonal, barrier contraceptive method
* Disease-free from prior nonbreast malignancies for at least 5 years before entry
* Adequate cardiac function( measured by baseline LVEF on MUGA or echocardiogram greater than or equal to the institution's lower limit of normal)

Exclusion criteria:

* Male
* Hormonal birth control
* The use of hormonal agents or raloxifene
* Active infection
* Pregnancy or breastfeeding
* Bilateral malignancy or a mass in the opposite breast suspicious for malignancy, unless there is biopsy proof that the mass is not malignant
* Previous therapy for breast cancer
* Nonmalignant systemic disease that would keep the patient from being given the treatment or would prevent long-term follow-up
* Active cardiac disease that would preclude the use of epirubicin and/or Taxol
* Significant abnormal peripheral nerve disease (greater than or equal to Grade 2)
* Any prior anthracycline or taxane-containing chemotherapy
* Use of any investigational agent within one month before enrollment
* Excisional biopsy of the breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76
Dates: Start 2001-11; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To determine the pathological response rate in tumors of patients with locally advanced breast cancer who receive 4 to 6 cycles of GET chemotherapy

SECONDARY OUTCOMES:
To determine the clinical response rate
to evaluate the toxicity of the GET combination
to determine feasibility of tissue collection and analysis of potential molecular and genetic correlates of response; to determine the 2-year survival and 2-year progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: John Hamm, MD, Study Chair — NSABP Foundation Inc; Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (1):
- NSABP Foundation, Inc., Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Hamm JT, Wilson JW, Rastogi P, Lembersky BC, Tseng GC, Song YK, Kim W, Robidoux A, Raymond JM, Kardinal CG, Shalaby IA, Ansari R, Paik S, Geyer CE, Wolmark N; NSABP Foundation Research Group. Gemcitabine/epirubicin/paclitaxel as neoadjuvant chemotherapy in locally advanced breast cancer: a phase II trial of the NSABP Foundation Research Group. Clin Breast Cancer. 2008 Jun;8(3):257-63. doi: 10.3816/CBC.2008.n.029. PMID 18650156